CLINICAL TRIAL: NCT01127243
Title: Do Women Prefer to Stay in Hospital Following Hysterectomy? A Randomised Trial of Day-case Versus Inpatient Laparoscopic Supracervical Hysterectomy
Brief Title: Day-case Versus Inpatient Laparoscopic Supracervical Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Jelena Kisic-Trope, Oslo university Hospital, Ullevål
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-08447a
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2009-06

CONDITIONS: Hysterectomy
Keywords: Hysterectomy; laparoscopy; day-case surgery; quality of life; Ambulatory Surgical Procedures
MeSH Terms: interventions — Ambulatory Surgical Procedures; Inosine Monophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- inpatient LSH (Active Comparator): LSH means laparoscopic supracervical hysterectomy
  Interventions: Procedure: inpatient LSH
- Day-case LSH (Experimental): LSH means laparoscopic supracervical hysterectomy
  Interventions: Procedure: day-case laparoscopic supracervical hysterectomy

INTERVENTIONS:
Procedure: day-case laparoscopic supracervical hysterectomy — patients discharged home the same day of the operation
  Other Names: day surgery, day-case, outpatient surgery
  Arms: Day-case LSH
Procedure: inpatient LSH — patients discharged home the day after the operation
  Other Names: inpatient, overnight stay
  Arms: inpatient LSH

SUMMARY:
The purpose of this study is to determine if women subjected to laparoscopic supracervical hysterectomy in a day-case setting would be less satisfied with the length of hospital stay when compared with women who had an overnight stay following their surgical procedure. The null hypothesis was that there was no difference in satisfaction with length of hospital stay.

DETAILED DESCRIPTION:
Objective: To determine whether women having day-case laparoscopic supracervical hysterectomy (LSH) are as satisfied with the length of stay in hospital as women who stay overnight following the procedure.

Design: randomised controlled trial (RCT).

Setting: Ulleval university hospital, Oslo, Norway.

Population: 49 women scheduled for LSH were enrolled and 45 patients completed the study (22 in the inpatient group and 23 in the day-case group).

Methods: Women were randomised to either day-case care or overnight hospital stay following a routine supracervical hysterectomy. The primary outcome measure was satisfaction with the length of stay in the hospital (measured on a 10-point visual analogue scale) and secondary measures were health-related quality of life (measured using the EuroQol EQ5D), anxiety (measured using the State-Trait Anxiety Inventory for Adults (STAI) and general questions about their experiences of having the operation. Readmissions, prolonged hospitalisations, complications and any contact with a health professional after discharge were also recorded. Measures were taken on the day of surgery (postoperatively), and on days 1, 2, 4 and 7 following surgery. The data were analysed based on an intention to treat.

ELIGIBILITY:
Inclusion Criteria:.

* women requiring a hysterectomy for benign conditions

Exclusion Criteria:

* previous history of cervical dysplasia, an abnormal smear test within the last two to three years,
* abnormal histology or cytology at endometrial sampling,
* a history of endometriosis,
* advanced endometriosis diagnosed intra-operatively,
* previous major abdominal or pelvic surgery (patients with previous caesarean section were considered as eligible),
* a mental disorder or somatic disease that would interfere with a normal recovery pattern such as substance dependence disorder,
* psychosis, or American Society of Anaesthesiologists (ASA) rating 3 and 4 patients, and
* inability to understand and execute oral and written Norwegian language.
* women were also excluded from the study if they did not have an adult carer (a relative or a friend) staying with them during the first night after discharge; or they were living or staying at a hotel more than an hour's drive from the hospital; and if they did not have access to a telephone.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
satisfaction with the length of stay in the hospital | on the 7th postoperative day
  satisfaction was measured on a 10-point visual analogue scale

SECONDARY OUTCOMES:
health-related quality of life | measured on days 1, 2, 4 and 7 following surgery
  health-related quality of life (measured using the EuroQol EQ5D), anxiety (measured using the State-Trait Anxiety Inventory for Adults (STAI) and general questions about their experiences of having the operation. Readmissions, prolonged hospitalisations, complications and any contact with a health professional after discharge were also recorded

CONTACTS AND LOCATIONS:
Overall Officials: Jelena Kisic-Trope, MD, Msc, Principal Investigator — Oslo University Hospital, Ullevål
Locations (1):
- Oslo University Hospital, Ullevål, Oslo, Oslo County, Norway